CLINICAL TRIAL: NCT05150925
Title: Immediate Mobilization Versus 2 Weeks Cast Immobilization After Distal Radius Fracture Treated With Volar Locking Plate - a Study Protocol for a Prospective, Randomized, Controlled Trial
Brief Title: Immediate Mobilization Versus 2 Weeks Cast Immobilization After Distal Radius Fracture Treated With Volar Locking Plate
Acronym: LIMPER-DRF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Kuopio University Hospital (Other); Jyväskylä Central Hospital (Other); Sundsvall Hospital (Other); Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Aleksi Reito, Associate professor, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21111
Record Dates: First submitted 2021-10-07; First posted 2021-12-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Distal Radius Fracture
Keywords: distal radius fracture; volar plating; surgery
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate mobilization after distal radius fracture treated with volar locking plate (Experimental)
  Interventions: Other: Immediate mobilization; Procedure: Volar plating
- 2 weeks cast immobilization after distal radius fracture treated with volar locking plate (Active Comparator)
  Interventions: Other: Cast treatment; Procedure: Volar plating

INTERVENTIONS:
Other: Cast treatment — Dorsal cast placed in OR
  Arms: 2 weeks cast immobilization after distal radius fracture treated with volar locking plate
Other: Immediate mobilization — Immediate mobilization postoperatively without casting
  Arms: Immediate mobilization after distal radius fracture treated with volar locking plate
Procedure: Volar plating — Volar plating of distal radius fracture

SUMMARY:
The aim of this study is to analyze total lenght of the sick leace and functional outcome (PRWE) at 2 months between 2 weeks casting and immediate mobilization following volar plating for a DRF.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled trial. The aim of this study will be to compare the early postoperative outcomes of the patients enrolled in the early mobilization with those patients in post-operative 2-week casting following volar plating for a DRF. Co-primary outcome in this study will be the total lenght of sick leave and Patient-Rated Wrist Evaluation (PRWE) 2 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Intra- or extra articular DRF (Colles, Smith, Volar barton)
* operative treatment justified

Exclusion Criteria:

* Refusal to participate in the study
* Open fracture with a severity greater than Gustilo grade 1
* Patient aged less than 18 or over 65
* Patient does not understand written or spoken guidance in local languages
* Pathological fracture
* Previous fracture in the same wrist or forearm in the last 10 years, that has led to impairment of function
* Ipsilateral fracture in upper extremity
* Associated fractures of the ulna (except fractures of the PSU)
* Polytrauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-02-10 (Actual); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Patient-rated wrist evaluation questionnaire | 2 months
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in daily activities. It ranges from 100 (worst) to 0 (best). It consists of 2 subscales. Pain subscale contains 5 items. Function subscale contains total 10 items which are further divided into 2 sections: specific activities (having 6 items) and usual activities.
Total lenght of the sick leave | 12 months
  Total number of days of work during the 1 year study period

SECONDARY OUTCOMES:
Patient-rated wrist evaluation questionnaire | 4 weeks
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in daily activities. It ranges from 100 (worst) to 0 (best). It consists of 2 subscales. Pain subscale contains 5 items. Function subscale contains total 10 items which are further divided into 2 sections: specific activities (having 6 items) and usual activities.
Patient-rated wrist evaluation questionnaire | 6 months
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in daily activities. It ranges from 100 (worst) to 0 (best). It consists of 2 subscales. Pain subscale contains 5 items. Function subscale contains total 10 items which are further divided into 2 sections: specific activities (having 6 items) and usual activities.
Patient-rated wrist evaluation questionnaire | 12 months
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in daily activities. It ranges from 100 (worst) to 0 (best). It consists of 2 subscales. Pain subscale contains 5 items. Function subscale contains total 10 items which are further divided into 2 sections: specific activities (having 6 items) and usual activities.
Return to work | 4 weeks
  Patient is asked if he or she has returned to the previous work. If no patient is asked is he or she Still on sick leave, partial sick leave or returned to other work.
Return to work | 2 months
  Patient is asked if he or she has returned to the previous work. If no patient is asked is he or she Still on sick leave, partial sick leave or returned to other work.
Return to work | 6 months
  Patient is asked if he or she has returned to the previous work. If no patient is asked is he or she Still on sick leave, partial sick leave or returned to other work.
Return to work | 12 months
  Patient is asked if he or she has returned to the previous work. If no patient is asked is he or she Still on sick leave, partial sick leave or returned to other work.
Complications | 4 weeks
  Any surgery related complication: wound dehiscence, deep infection, flexor tendon rupture, nerve injury, mechanical complications, nonunion, malunion, complex regional pain syndrome
Complications | 2 months
  Any surgery related complication: wound dehiscence, deep infection, flexor tendon rupture, nerve injury, mechanical complications, nonunion, malunion, complex regional pain syndrome
Complications | 6 months
  Any surgery related complication: wound dehiscence, deep infection, flexor tendon rupture, nerve injury, mechanical complications, nonunion, malunion, complex regional pain syndrome
Complications | 12 months
  Any surgery related complication: wound dehiscence, deep infection, flexor tendon rupture, nerve injury, mechanical complications, nonunion, malunion, complex regional pain syndrome
Self-perceived working ability | 4 weeks
  Patient is asked to rate his os her working ability using two scales: NRS from 0 (fully disabled) to 10 (best capability) and ordinally (fully capable, partially capable, fully disabled).
Self-perceived working ability | 2 months
  Patient is asked to rate his os her working ability using two scales: NRS from 0 (fully disabled) to 10 (best capability) and ordinally (fully capable, partially capable, fully disabled).
Self-perceived working ability | 6 months
  Patient is asked to rate his os her working ability using two scales: NRS from 0 (fully disabled) to 10 (best capability) and ordinally (fully capable, partially capable, fully disabled).
Self-perceived working ability | 12 months
  Patient is asked to rate his os her working ability using two scales: NRS from 0 (fully disabled) to 10 (best capability) and ordinally (fully capable, partially capable, fully disabled).
Visual analogue pain scale | 4 weeks
  Overall pain during last 7 days in a scale from 0 to 100 (worst)
Visual analogue pain scale | 2 months
  Overall pain during last 7 days in a scale from 0 to 100 (worst)
Visual analogue pain scale | 6 months
  Overall pain during last 7 days in a scale from 0 to 100 (worst)
Visual analogue pain scale | 12 months
  Overall pain during last 7 days in a scale from 0 to 100 (worst)
Patient-acceptable symptom state | 2 months
  Patient satisfaction will be measured using the patient-acceptable symptom state (PASS).The questionnaires will include the following questions: Would you be willing to take the same treatment again if the treatment result was as it is now? (Yes/No) Considering all the different ways your injury is affecting you, if you would remain in this state, do you feel that your current state is satisfactory (Yes/No)?
Patient-acceptable symptom state | 6 months
  Patient satisfaction will be measured using the patient-acceptable symptom state (PASS).The questionnaires will include the following questions: Would you be willing to take the same treatment again if the treatment result was as it is now? (Yes/No) Considering all the different ways your injury is affecting you, if you would remain in this state, do you feel that your current state is satisfactory (Yes/No)?
Patient-acceptable symptom state | 12 months
  Patient satisfaction will be measured using the patient-acceptable symptom state (PASS).The questionnaires will include the following questions: Would you be willing to take the same treatment again if the treatment result was as it is now? (Yes/No) Considering all the different ways your injury is affecting you, if you would remain in this state, do you feel that your current state is satisfactory (Yes/No)?
Work capacity | 4 weeks
  The participants will be asked to rate their working capacity on a numerical scale from 0 to 10, with "0" being not able to work at all and "10" being the ability to work at its best.
Work capacity | 2 months
  The participants will be asked to rate their working capacity on a numerical scale from 0 to 10, with "0" being not able to work at all and "10" being the ability to work at its best.
Work capacity | 6 months
  The participants will be asked to rate their working capacity on a numerical scale from 0 to 10, with "0" being not able to work at all and "10" being the ability to work at its best.
Work capacity | 12 months
  The participants will be asked to rate their working capacity on a numerical scale from 0 to 10, with "0" being not able to work at all and "10" being the ability to work at its best.

OTHER OUTCOMES:
Patient activity | 4 weeks
  Patient activity measured with triaxial wrist accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Aleksi Reito, Study Director — Tampere University Hospital; Laura Kärnä, MD, Principal Investigator — Tampere University Hospital
Locations (5):
- Finland (3):
  - Teemu Karjalainen, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Laura Kärnä, Tampere
- Sweden (2):
  - Danderyds Sjukhus, Danderyd
  - Sundsvalls sjukhuset, Sundsvall

IPD SHARING:
Plan to Share IPD: Yes
Data is available on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After the study has been completed and for 10 years after.
Access Criteria: On reasonable request and research plan for IPD use should be provided.

REFERENCES:
- [Derived] Karna L, Launonen AP, Karjalainen T, Luokkala T, Ponkilainen V, Halonen L, Helminen M, Mattila VM, Reito A. LIMPER trials: immediate mobilisation versus 2-week cast immobilisation after distal radius fracture treated with volar locking plate - a study protocol for a prospective, randomised, controlled trial. BMJ Open. 2022 Nov 11;12(11):e064440. doi: 10.1136/bmjopen-2022-064440. PMID 36368761

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT05150925/SAP_000.pdf